CLINICAL TRIAL: NCT07295249
Title: Asthma Health Literacy Scale for Children (AHLSC) (Aged 8-12): A Scale Development Study
Brief Title: Asthma Health Literacy Scale for Children (AHLSC) (Aged 8-12)
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Fatma Yeşil, Lecturer Dr, University of Yalova
Other Study IDs: YU-TSHMYO-FY-01
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Asthma (Diagnosis); Children; Health Literacy; Scale Reliability Validity
Keywords: Asthma; health literacy; child; scale development; nursing
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A Scale Development Study: The research was conducted with 196 children aged 8-12 diagnosed with asthma. Participants were reached via an online survey form. Study data were collected using a "Participant Information Form" and the "Asthma Health Literacy Scale for Children (ASOYÖ) (8-12 years)," filled out by the children themselves.
  Interventions: Other: Asthma Health Literacy Scale for Children (AHLSC) (Aged 8-12): A Scale Development Study

INTERVENTIONS:
Other: Asthma Health Literacy Scale for Children (AHLSC) (Aged 8-12): A Scale Development Study — This study was conducted using a methodological design to develop and test the psychometric properties of the "Asthma Health Literacy Scale for Children (ASOYÖ)" for children aged 8-12.

SUMMARY:
Asthma Health Literacy Scale for Children (AHLCS) (Ages 8-12): A Scale Development Study

Objective: This study will be conducted using a methodological design to develop and examine the psychometric properties of the Asthma Health Literacy Scale for Children (AHLCS) for children aged 8-12 years.

DETAILED DESCRIPTION:
This research was conducted to develop the Asthma Health Literacy Scale for children and to test its psychometric properties. The research is a methodological scale development study.

A review of the national and international literature revealed no studies measuring the health literacy level of children with asthma, indicating a significant gap in this area. It is therefore thought that the developed scale will fill an important gap. With this understanding, children's information level requirements regarding asthma can be identified; specific initiatives can be planned to meet the identified requirements of children; and, accordingly, children's asthma health literacy information level regarding asthma can be measured.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with asthma for at least one year.
* Not having any mental and/or physical health problems that would prevent communication.
* Agreeing to participate in the research.
* Parental consent obtained.
* Being between the ages of 8-12.

Exclusion Criteria:

* Children who filled out the data forms incompletely.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children diagnosed with asthma aged 8-12
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Asthma Health Literacy Scale for Children (AHLSC) (Aged 8-12) | 2 months
  The initial form of the scale was developed with 28 items; as a result of validity and reliability analyses, a structure consisting of 19 items and 2 sub-dimensions was obtained.
  The scale is 4-point Likert type, and response options are 1=Never, 2=Sometimes, 3=Often, 4=Always. Each item is scored between 1-4, and the minimum score obtainable from the scale is 19, and the maximum is 76. As the total score increases, the asthma health literacy level of children diagnosed with asthma increases. There are no reverse-scored items in the scale.
  The developed scale is a valid and reliable tool for assessing the health literacy levels regarding asthma in children aged 8-12.Participants were reached via an online survey form. Study data were collected using a "Asthma Health Literacy Scale for Children" filled out by the children themselves.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda CAN, Assoc Prof, Study Chair — University of Yalova
Locations (1):
- Emel Avçin, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No